CLINICAL TRIAL: NCT05656313
Title: Feature Supporting Multitasking of Visual and Acoustical Objects
Brief Title: PRINCE22 System Complete Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SRF-2391
Record Dates: First submitted 2022-11-16; First posted 2022-12-19 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2022-12

CONDITIONS: Hearing Loss, Bilateral; Hearing Loss, Unilateral
MeSH Terms: conditions — Hearing Loss, Bilateral; Hearing Loss, Unilateral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrow reference beamformer (Experimental)
  Interventions: Device: Measures of speech intelligibility in a noisy situation with speech from the side and from behind (measured with CC-OLSA Test); Device: Measures of the subjective speech recognition threshold in a noisy situation with speech from the side and from behind (measured with HEISS test); Device: Ability to multitask in the auditory and visual domains in noisy situation with speech from the side and from behind (Multitask test); Device: Measure of subjective speech intelligibility and listening effort in noisy situation with speech from the side and from behind (subjective assessment; 100-point scale)
- Novel beamformer approach (Active Comparator)
  Interventions: Device: Measures of speech intelligibility in a noisy situation with speech from the side and from behind (measured with CC-OLSA Test); Device: Measures of the subjective speech recognition threshold in a noisy situation with speech from the side and from behind (measured with HEISS test); Device: Ability to multitask in the auditory and visual domains in noisy situation with speech from the side and from behind (Multitask test); Device: Measure of subjective speech intelligibility and listening effort in noisy situation with speech from the side and from behind (subjective assessment; 100-point scale)

INTERVENTIONS:
Device: Measures of speech intelligibility in a noisy situation with speech from the side and from behind (measured with CC-OLSA Test) — The Concurrent OLSA test (CC-OLSA) is a speech recognition test with three turn-taking talkers presenting sentences of the Oldenburg sentences test at fixed signal-to-noise ratios.
  CC-OLSA is the only one-talker-at-a-time speech test that is sensitive at the desired SNR and uses sentences with an intelligibility function with slopes of 10-17 %/dB.
Device: Measures of the subjective speech recognition threshold in a noisy situation with speech from the side and from behind (measured with HEISS test) — The measure of the subjective speech recognition threshold is an alternative procedure to evaluate the subjective speech intelligibility in different listening conditions. The subjective speech recognition threshold is defined as the speech presentation level of running speech needed to just follow conversation. Subjects have to adjust the presentation level of speech so that they are just able to understand the speech, using a slider on a touch screen. This adjustment is repeated 10 times. Each adjustment results in a value for the subjective speech recognition threshold in dB SNR. The outcome measure is the mean value of the 10 repetitions. The HEISS-Test will be repeated four times for the secondary objective: test for 2 test conditions (Reference, novel approach) against 2 target directions (better ear side, back).
Device: Ability to multitask in the auditory and visual domains in noisy situation with speech from the side and from behind (Multitask test) — This test uses a dual-task-paradigm assessing vigilance for auditory and visual triggers concurrently. The primary task is to listen to a novel (Harry Potter) and respond on two trigger words by pressing the appropriate button (one in each hand). The secondary task is to observe a monitor showing a sequence of random signs and respond on a target sign by pressing both buttons. The test includes at least 100 triggers (50 auditory, 50 visual) and takes 10 minutes per condition (side vs. back; novel approach vs. reference; 40 minutes in total). The multitask test will be repeated four times for the secondary objective: 2 conditions (Refrence, novel approach) against 2 target directions (better ear side, back). Following data are provided from each multitask Test measure: (1) subjective rating of the perceived ability to perform the visual and the auditory test simultaneously. (2) reaction times to auditory and visual tasks, and (3) accuracy.
Device: Measure of subjective speech intelligibility and listening effort in noisy situation with speech from the side and from behind (subjective assessment; 100-point scale) — In addition to the tests mentioned above a subjective assessment will be used to determine the subjective perception as this measure is often a good indication for clinical relevance.
  For this purpose, the same speech material as used in the HEISS-test is presented by a loudspeaker in the same noisy environment as in the other three tests. The subjects rate his/her perception of the presented speech using a questionnaire on the dimensions "listen effort and speech intelligibility". The subject will rate his perception on the 100 point scale with pencils with different colors to get either absolute and relative ratings.
  The subjective assessment will be repeated four times for the secondary objective: 2 test conditions (Rference and novel approach) against 2 target directions (better ear side, back). Following data are provided from assessment: rating on a 100-point scale per condition and per dimension.

SUMMARY:
The investigation proposes to compare a narrow reference beamformer to a novel beamformer approach, when the talker is not in front of the hearing aid user and in the presence of background noise. The beamformer effect will be determined in terms of speech intelligibility, listening effort and ability to multitask when the talkers are located on the side or in the back.

ELIGIBILITY:
Inclusion Criteria:

* Experienced (minimum use duration 6 months)
* Adult (minimum age: 18 years) hearing aid users,
* Written and spoken German,
* Ability to understand instruction,
* Ability to perform tests successfully
* Ability to describe listening experiences,
* Ability to attend to the appointments,
* Healthy outer ear,
* Moderat to severe Hearing
* Informed consent as documented by signature.

Exclusion Criteria:

* Clinical contraindications deformity of the ear (closed ear canal or absence of pinna),
* Known hypersensitivity or allergy,
* Not willing to wear the hearing aid,
* Fluctuating hearing that could influence the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Difference in speech intelligibility between the reference beamformer and the novel beamformer approach (percentage of correct responses in word recognition) in a noisy situation with speech from the side and from behind. | 4 weeks
  Two directional conditions (better ear side, back) and two beamformer conditions (Novel approach: SpeechSensor, Reference: StereoZoom) are tested (test and retest, eight measurements in total).

SECONDARY OUTCOMES:
Difference in speech recognition threshold between the reference beamformer and the novel (mean value of 10 repetitions). | 4 weeks
  Subjects have to adjust the presentation level of speech so that they are just able to understand the speech, using a slider on a touch screen. This adjustment is repeated 10 times. Each adjustment results in a value for the subjective speech recognition threshold in dB signal-to-noise ratio.
Difference in multitasking ability between the reference beamformer and the novel (1. Respond on two trigger words / 2. Respond on a target sign). | 4 weeks
  This test uses a dual-task-paradigm assessing vigilance for auditory and visual triggers concurrently. The primary task is to listen to a novel (Harry Potter) and respond on two trigger words by pressing the appropriate button (one in each hand). The secondary task is to observe a monitor showing a sequence of random signs and respond on a target sign by pressing both buttons. The test includes at least 100 triggers (50 auditory, 50 visual) and takes 10 minutes per condition (side vs. back; SpeechSensor vs. StereoZoom; 40 minutes in total).
Difference in subjective speech intelligibility between the reference beamformer and the novel (subjects rate his/her perception of the presented speech). | 4 weeks
  The subjects rate his/her perception of the presented speech using a questionnaire on the dimensions "listen effort and speech intelligibility". The subject will rate his perception on the 100 point scale with pencils with different colors to get either absolute and relative ratings. The subjective assessment will be repeated four times for the secondary objective: 2 test conditions (StereoZoom and SpeechSensor) against 2 target directions (better ear side, back). Following data are provided from assessment: rating on a 100-point scale per condition and per dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Latzel, Study Director — Sonova AG
Locations (1):
- Hörzentrum Oldenburg gGmbH, Oldenburg, Lower Saxony, Germany